CLINICAL TRIAL: NCT07015970
Title: Suivi en Vie Réelle de l'Activité Physique de Patients Présentant un Diabète de Type 1 Sportifs Equipés d'Une Pompe à Insuline Avec Délivrance Automatisée d'Insuline
Brief Title: Real-life Follow-up of the Physical Activity in Type 1 Diabetes Participants Equipped With an Insulin Pump With Hybrid Closed Loop
Acronym: RAPPID
Status: Completed | Type: Observational
Sponsor: ISIS Diabete Service (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A01901-44
Record Dates: First submitted 2025-05-23; First posted 2025-06-11 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus Type 1; Glucose Metabolism Disorder; Glycemic Control for Diabetes Mellitus; Fear of Hypoglycemia; Treatment Satisfaction; Quality of Life; Hypoglycaemia
Keywords: Automated insulin delivery; Exercice; Diabetes Mellitus, Type 1; Hypoglycemia; Glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Adults with type 1 diabetes mellitus using AID and engaging in regular physical activity
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention

SUMMARY:
This is a non-interventional, prospective, multi-site study conducted in France among adults with type 1 diabetes mellitus using automated insulin delivery (AID) systems and engaging in at least two exercise sessions per week, each lasting at least 30 minutes. The main objective of this study is to describe the glycemic control of athletic participants with type 1 diabetes mellitus who use an insulin pump with AID and engage in physical exercise under real-life conditions.

Two physician data collection time points are planned: the first occurs at baseline and includes demographic and clinical data, glycemic control during the month preceding inclusion, diabetes management, and information on usual physical exercise (duration, type, sport practiced, competition participation, and adherence to a specific diet). The second occurs at 1-month follow-up and involves downloading insulin pump and glucose sensor data, covering the period from 15 days before the first reported exercise session to 15 days after the last session.

During the 1-month study period, participants will complete a paper logbook after each exercise session to document information such as the type of exercise, self-reported intensity using the modified Borg scale and the WHO physical activity intensity scale, duration, system adjustments, dietary intake, occurrence of hypoglycemia and associated symptoms, snacks consumed, and treatments administered for hypoglycemia.

DETAILED DESCRIPTION:
Three hybrid closed-loop systems dedicated to the automated management of type 1 diabetes are currently available in France: the Minimed 780G paired with the Guardian 4 continuous glucose monitoring system, Control-IQ, and mylife CamAPS-FX. Stratification will be performed based on the type of pump used by participants at the time of inclusion, at the national level, in order to obtain groups balanced in size.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants with diabetes mellitus type 1
* User for at least 3 months of one the three automated insulin delivery systems available in France at the time of the study (Minimed 780G pump + Guardian 4 sensor + PID-IFB algorithm; or T:Slim X2 pump + Dexcom G6 sensor + Control-IQ algorithm; or mylife Ypsopump + Dexcom G6 sensor + CamAPS FX app)
* Engaged in regular physical activity as part of daily life (at least 2 structured sessions per week, each lasting more than 30 minutes)
* Able to download data from the pump
* Willing and able to complete the physical activity log and self-questionnaires in French
* Having received the information sheet and given their oral consent (non-opposition) to participate in the study and for their data processing

Exclusion Criteria:

* Participants currently enrolled in a clinical trial
* Pregnancy or breastfeeding women or women planning a pregnancy during the study
* Adults under legal protection (guardianship, curatorship, or judicial safeguard)
* Participants with decompensated retinopathy
* Participants with decompensated cardiac disease
* History of severe hypoglycemia during physical activity in the past 6 months
* Participants with unresolved diabetic foot trophic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be recruited by four specialized tertiary diabetes care centers (Vandœuvre-lès-Nancy, Strasbourg, Caen, and Mainvilliers).
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Time Below Range | One month
  Percentage of time spent with glucose <70 mg/dL and <54 mg/dL before the exercise (within 2 hours prior), during exercise, during early recovery (within 3 hours after exercise), late recovery (from 3 hours after exercise to 8:00 a.m. the following day or until the next pre-exercise window, if closely), and during non-exercise periods

SECONDARY OUTCOMES:
Time-in-Range | One month
  Percentage of time spent in target glucose range 70-180 mg/dL before the exercise (within 2 hours prior), during exercise, during early recovery (within 3 hours after exercise), late recovery (from 3 hours after exercise to 8:00 a.m. the following day or until the next pre-exercise window, if closely), and during non-exercise periods
Time Above Range | One month
  Percentage of time spent with glucose >180 mg/dL and >250 mg/dL before the exercise (within 2 hours prior), during exercise, during early recovery (within 3 hours after exercise), late recovery (from 3 hours after exercise to 8:00 a.m. the following day or until the next pre-exercise window, if closely), and during non-exercise periods
Ajustement Practices | One month
  Reported by participants and available from insulin pump data before, during and after exercise sessions
ADDQoL questionnaire | At inclusion
  Self-administered questionnaire: Audit of Diabetes-Dependent Quality of Life (ADDQoL), including three scores:
  The first concerns the perceived quality of life, with 7 items ranging from "extremely poor" to "excellent." Total scores range from -3 to +3, with higher scores reflecting better quality of life.
  The second concerns the quality of life if the participant did not have diabetes, with 5 items ranging from "much better" to "worse." Total scores range from -3 to +1, with higher scores indicating that life would be significantly worse without diabetes.
  The third concerns the impact of diabetes on specific life domains, with 19 items ranging from "much better" to "worse," combined with the personal importance of each domain, rated from 0 (not at all important) to 3 (very important). The resulting weighted ADDQoL scores range from -9 to +3, with higher scores reflecting the maximum positive impact of diabetes.
DTSQs questionnaire | At inclusion
  Self-administered questionnaire: Diabetes Treatment Satisfaction Questionnaire (DTSQs), consisting of 8 items ranging from 0 to 6. Total scores range from 0 to 36, with higher scores indicating better treatment satisfaction.
HFS-II questionnaire | At inclusion
  Self-administered questionnaire Hypoglycemia Fear Survey II (HFS-II) composed of two subscales: a Behaviour score and a Worry score, each consisting of 4 items rated from 0 (never) to 4 (almost always). Total scores range from 0 to 16 with higher scores reflecting greater behavioural or emotional impact.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno GUERCI, Professor, MD, PhD, Principal Investigator — CHRU Nancy and University of Lorraine, Nancy, france
Locations (4):
- France (4):
  - CHU of Caen, Caen
  - Institute of Diabetology, Mainvilliers
  - CHRU of Nancy, Nancy
  - University Hospitals of Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No
In accordance with the General Data Protection Regulation and French data protection law, the presentation of the results derived from data processing shall under no circumstances allow the direct or indirect identification of individuals participating in the research.
  In the event of publication of the research findings in a scientific journal, access to the data by an independent expert - including one appointed by a scientific publisher - shall only be granted through the interface provided or designated by the Data Controller, solely for the purpose of verifying or reproducing the analyses, and exclusively under the conditions defined for secure consultation and data handling.

REFERENCES:
- [Result] Joubert M, Meyer L, Bekka S, Rakotoarisoa L, Scheyer N, Dreves B, Guerci B. Hypoglycemia incidence and behavioural adjustments during free-living unstructured physical activity in adults with type 1 diabetes using AID systems: Results from the RAPPID study. Diabetes Obes Metab. 2025 Dec;27(12):7221-7231. doi: 10.1111/dom.70122. Epub 2025 Sep 9. PMID 40926369